CLINICAL TRIAL: NCT06163781
Title: Appropriate Use of Blood Cultures in the Emergency Department Through Machine Learning: a Randomized Controlled Trial
Brief Title: Appropriate Use of Blood Cultures in the Emergency Department Through Machine Learning
Acronym: ABC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Prabath W.B. Nanayakkara, MD, PhD, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL81971.000.22
Record Dates: First submitted 2023-10-12; First posted 2023-12-11 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Artificial Intelligence; Machine Learning; Microbiology; Emergency Service, Hospital; Randomized Controlled Trial
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood culture taken based on machine learning tool (Experimental)
  Interventions: Device: Blood culture prediction tool
- Blood culture taken based on the treating physician (No Intervention)

INTERVENTIONS:
Device: Blood culture prediction tool — Machine learning based predicition tool
  Arms: Blood culture taken based on machine learning tool

SUMMARY:
The goal of this clinical trial is to study whether the use of our blood culture prediction tool is non-inferior to current practice and if it can improve certain outcomes in all adult patients presenting to the emergency department with a clinical indication for a blood culture analysis (according to the treating physician). The primary endpoint is 30-day mortality. Key secondary outcomes are:

* hospital admission rates
* in-hospital mortality
* hospital length-of-stay. In the intervention group, the physician will follow the advice of our blood culture prediction tool.

In the comparison group all patients will undergo a blood culture analysis.

DETAILED DESCRIPTION:
Rationale: The overuse of blood cultures in emergency departments leads to low yields and high numbers of contaminated cultures, which is associated with increased diagnostics, antibiotic usage, prolonged hospitalisation, and mortality. Ideally, blood cultures would only be performed in patients with a high risk for a positive culture. The investigators have developed a machine learning model to predict the outcome of blood cultures in the ED. Retrospective and prospective validation of the tool in various settings show that it can be used to reduce the number of blood culture analyses by at least 30% and help avoid the hidden costs of contaminated cultures.

Objective: This study aims to investigate whether the use of our blood culture prediction tool is non-inferior to current practice and if it can improve certain outcomes.

Study design: A randomized controlled non-inferiority trial. Study population: All adult patients presenting to the emergency department with a clinical indication for a blood culture analysis (according to the treating physician).

Intervention: In the control group, all patients will undergo a blood culture analysis. In the intervention group, the physician will follow the advice of our blood culture prediction tool. If the chance of a positive blood culture is < 5%, the blood culture analysis will be cancelled and the sample destroyed. If the change of a positive blood culture is > 5%, the blood culture analysis will be performed as usual.

Main study parameters/endpoints: The primary endpoint is 30-day mortality, for which the investigators aim to show non-inferiority. Key secondary outcomes, for which the investigators also aim to show non-inferiority, are hospital admission rates, in-hospital mortality, and hospital length-of-stay.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Have a clinical indication for a blood culture analysis (according to the treating physician)
* Have sufficient data recorded (laboratory results and vital sign measurements) for a prediction to be made (at least 20% of the needed parameters)

Exclusion Criteria:

* Central Venous Line (CVL) or Peripherally Inserted Central Catheter (PICC) in situ
* Neutrophil count < 0.5 * 109/L
* Candidemia or S. aureus bacteraemia in the past 3 months.
* Most likely diagnosis of endocarditis/spondylodiscitis/infected prosthetic material
* Pregnant or breastfeeding patients
* Not capable of giving informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7584 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
30-day mortality | 30 days

SECONDARY OUTCOMES:
hospital admission rates | 1 day
in-hospital mortality | 90 days
hospital length-of-stay | 90 days

OTHER OUTCOMES:
30-day readmission rates | 30 days
Length of stay in the ED in hours | 2 days
Percentage of blood cultures avoided in the intervention group | 90 days
90 day mortality | 90 days
Number of blood cultures on each day of hospital stay (in admitted patients) | 90 days
Percentage of positive blood cultures in each group | 90 days
Total number of laboratory- and microbiology tests in the ED | 2 days
Total number of laboratory- and microbiology test on each day of hospital stay (in admitted patients) | 90 days
Percentage of patients receiving antibiotics in the ED | 2 days
Duration of antibiotic therapy | 90 days
Types of antibiotics given in the ED | 2 days
Model performance (AUC) during the trial | 3 years
Model performance in subgroup of Immunocompromised patients (triple immunosuppressive therapy) | 3 years
Model performance in subgroup of transplanted patients | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC - location AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
: Participant data underlying the results of this study can be shared. The data can be requested following publication of this work. The data can be shared with researchers who provide a methodologically sound proposal, which is allowed under our local privacy regulations. Proposals should be directed to the corresponding author and requestors will need to sign a data access agreement.

REFERENCES:
- [Result] Boerman AW, Schinkel M, Meijerink L, van den Ende ES, Pladet LC, Scholtemeijer MG, Zeeuw J, van der Zaag AY, Minderhoud TC, Elbers PWG, Wiersinga WJ, de Jonge R, Kramer MH, Nanayakkara PWB. Using machine learning to predict blood culture outcomes in the emergency department: a single-centre, retrospective, observational study. BMJ Open. 2022 Jan 4;12(1):e053332. doi: 10.1136/bmjopen-2021-053332. PMID 34983764
- [Result] Schinkel M, Boerman AW, Bennis FC, Minderhoud TC, Lie M, Peters-Sengers H, Holleman F, Schade RP, de Jonge R, Wiersinga WJ, Nanayakkara PWB. Diagnostic stewardship for blood cultures in the emergency department: A multicenter validation and prospective evaluation of a machine learning prediction tool. EBioMedicine. 2022 Aug;82:104176. doi: 10.1016/j.ebiom.2022.104176. Epub 2022 Jul 16. PMID 35853298
- [Derived] van der Zaag AY, Bhagirath SC, Boerman AW, Schinkel M, Paranjape K, Azijli K, Ridderikhof ML, Lie M, Lissenberg-Witte B, Schade R, Wiersinga J, de Jonge R, Nanayakkara PWB. Appropriate use of blood cultures in the emergency department through machine learning (ABC): study protocol for a randomised controlled non-inferiority trial. BMJ Open. 2024 May 31;14(5):e084053. doi: 10.1136/bmjopen-2024-084053. PMID 38821574